CLINICAL TRIAL: NCT05848778
Title: Novel Non-invasive Therapy to Drive Robust and Sustained Peripheral Nerve Regeneration
Brief Title: Non-invasive Therapy to Drive Nerve Regeneration
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Royal Alexandra Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00128891
Record Dates: First submitted 2023-04-05; First posted 2023-05-08 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Peripheral Nerve Injuries
MeSH Terms: conditions — Peripheral Nerve Injuries

STUDY DESIGN:
Intervention Model Description: This study will investigate AIH's potential to condition and promote enhanced repair in a Phase I randomized control trial (RCT) of carpal tunnel syndrome (CTS) associated with severe median nerve compression/injury. We predict AIH will have better outcomes than current ES strategies and we aim to non-invasively condition/prime the IRP in compressed nerves by AIH treatment prior to nerve decompression and/or post-nerve decompression.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acute Intermittent Hypoxia (Active Comparator): Patients with hand weakness and numbness secondary to median nerve entrapment and scheduled for carpal tunnel release surgery will be randomly assigned to receive acute intermittent hypoxia
  Interventions: Device: Acute Intermittent Hypoxia
- Normoxia control (Placebo Comparator): Patients with hand weakness and numbness secondary to median nerve entrapment and scheduled for carpal tunnel release surgery will be randomly assigned to receive normoxia
  Interventions: Device: Normoxia

INTERVENTIONS:
Device: Acute Intermittent Hypoxia — The acute intermittent hypoxia protocol will consist of 15 cycles of 1.5 min of inspiring ambient air (21% O2) alternating with 1.5 min of hypoxic air (9% O2)
  Arms: Acute Intermittent Hypoxia
Device: Normoxia — The normoxia protocol will consist of 15 cycles of 3 min of inspiring ambient air (21% O2)
  Arms: Normoxia control

SUMMARY:
Peripheral nerve injuries are common and often associated with poor outcomes including incomplete repair, debilitating pain states and compromised function. Although nerve regeneration can be enhanced by brief electrical nerve stimulation at the time of or before surgical repair in rodents and humans, this approach is invasive. Acute intermittent hypoxia, breathing alternate cycles of regular air and air with ~50% normal oxygen levels (11% O2) is an emerging, promising non-invasive therapy promoting respiratory and non-respiratory muscle function in spinal cord injured rats and humans. Because the entire body is exposed to this therapy, it has the potential to globally impact the nervous system beyond just controlling respiratory and leg function in spinal cord injured patients. Thus, the investigators hypothesized that an acute intermittent hypoxia paradigm similar to that used for spinal cord repair will improve peripheral nerve repair in a manner akin to electrical stimulation, including its impact on expression of regeneration-associated proteins - a predictor of nerve growth states. In recent studies the investigators found this to be the case and now propose to continue these promising studies by performing a pilot clinical trial evaluating this form of treatment on patients with compromised hand function due to severe carpal tunnel syndrome. The goal is to improve nerve repair outcomes in the least invasive and optimal manner.

DETAILED DESCRIPTION:
Peripheral nerve injuries are frequent and disabling, often with irreversible consequences. Injured sensory and motor neurons induce cellular and molecular events we refer to as the intrinsic repair program, linked to their regeneration capacity. Regrettably, regeneration of these nerves is challenging. Issues include whether the intrinsic repair program is robust enough, or is sustained long enough, to ensure repair over long distances. This can result in incomplete repair and/or pain states. The investigators will exploit acute intermittent hypoxia (intermittent periods of reduced oxygen), a novel treatment to condition/prime peripheral nerves and induce an enhanced intrinsic repair program. Acute intermittent hypoxia is non-invasive and has a systemic effect which is a major advantage in cases where there are multiple nerve injured in a widespread distribution, as opposed to electrical stimulation that only impacts the individual nerve stimulated. However, the full potential of acute intermittent hypoxia in nerve repair remains unknown. This will be a Phase I randomized control trial of carpal tunnel syndrome associated with severe median nerve compression/injury. This is designed to test the hypothesis that acute intermittent hypoxia before and/or after nerve decompression will result in more effective nerve regeneration and restoration of function.

Methods:

Using a double blinded randomized controlled trial design, we will recruit 80 adult patients (50% male; 50% female) >18 yrs old with severe carpal tunnel syndrome.

Statistical analysis:

Distribution of the outcome data will be analyzed using the Shapiro-Wilk test. For parameters that are normally distributed, differences between the groups will be compared using 2-way analysis of variance (ANOVA) with time and treatment allocation being the independent factors. When a statistically significant difference (p<0.05) is found, post hoc testing will be done using the Tukey test. For data that is not normally distribution, the Kruskal-Wallis test will be used instead, followed by post hoc analysis with Dunn's test when a significant difference is found. Sample size estimation - Assuming that AIH has a modest treatment effect size of 0.6 compared to the Normoxia control group, with type I error set at 0.05 and type II error at 0.80, appropriately 20 subjects are needed in each group to provide sufficient power for the study.

ELIGIBILITY:
Inclusion Criteria:

i) sensory impairments including numbness and pain; ii) nocturnal awakening by these symptoms; iii) weakness and wasting of the thenar musculature and, iv) loss of hand dexterity. v) Motor unit loss greater than 2 SD below the mean for the age group

Exclusion Criteria:

i) Chronic lung or cardiac disease ii) Other nerve disorders, previous carpal tunnel release or systemic illness including diabetes

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Motor unit number estimation | At 3, 6 and 12 months compared to baseline
  The number of motor units in the median innervated thenar muscles.

SECONDARY OUTCOMES:
Two point discrimination | At 3, 6 and 12 months compared to baseline
  Testing the A-beta sensory fibers using the Dellon-MacKinnon Disk
Fine touch sensation | At 3, 6 and 12 months compared to baseline
  Testing the A-beta fibers using Semmes-Weinstein monofilaments
Quantitative sensory testing | At 3, 6 and 12 months compared to baseline
  Cold threshold (A-beta fibers) and pain threshold (C fibers) using CASE IV quantitative sensory testing equipment
Boston Carpal Tunnel Symptom Severity | At 3, 6 and 12 months compared to baseline
  Self administered questionnaire
Moberg Pick-up Test | At 3, 6 and 12 months compared to baseline
  To measure hand dexterity and functional performance

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No